CLINICAL TRIAL: NCT01895816
Title: Phase 3 of Study on Effects of New Herbal Mixture on Men Infertility
Brief Title: Herbal Tonic Fertile Supplement(ZO2C5)
Acronym: (ZO2C5)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arash Khaki (Other)
Collaborators: Islamic Azad University of Tabriz (Other); Tabriz University (Other)
Responsible Party: Sponsor-Investigator, Arash Khaki, Clinical professor. Women's Reproductive Health Research Center, Tabriz University of Medical Sciences, Tabriz, Iran., Islamic Azad University of Tabriz
Organization: Islamic Azad University of Tabriz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: WRHRC-9026
Record Dates: First submitted 2012-09-12; First posted 2013-07-11 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Male Infertility
Keywords: male infertility,oligo spermia
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fertility coated tablet (Experimental): 700 mg fertility coated tablet containing 8 herbal powders by mouth every 12 hours for 180 days
  Interventions: Dietary Supplement: coated tablet

INTERVENTIONS:
Dietary Supplement: coated tablet — this supplement contains 700 mg of 8 natural herbals: Citrus & ZINGIBER OFFICINALE & Onion & Ocimum basilicum & Cinnamomum zelanicum & Citrullus lanatus & Citrullus vulgaris & Daucus carota
  Other Names: Dietry supplement

SUMMARY:
The purpose of this study is to determine whether the effect of mixed herbals drug (citrus, citrolus vol, lan, carrot seed, zingiber, onion, basil, cinnamon) administration on male infertility: oligospermia

DETAILED DESCRIPTION:
In the last few years, a marked decrease in the quality of semen has been reported. Infertility is one of the major health problems in 10 to 15% of couples' lives; from which approximately 50% of couple's infertility is due to Male factors. The aim of the present study was to evaluate an herbal mixed effects on spermatogenesis and the normal production of sperm. Researchers have reported that using antioxidants and vitamins A, B, C, E, flavonoids, Sulfur compounds, terpenoids and phenolic compounds in the daily diet can protect sperm. In this study the investigators aimed to assess synergistic effect of these herbal compounds in male Infertility. 700 mg tablet for 180 consequence days/daily will be advising, for 40 patients semen samples in 1th and 180 day after treatment will take, in andrology lab according WHO method:samples put into 2 mL of medium (Hams F10) containing 0.5% bovine serum albumin. After 5 min incubation at 37oC (with 5% CO), the sperm samples were determined using the standard haemocytometric method, and sperm motility was analyzed by microscope (Olympus IX70) at 10 field and reported as the mean of motile sperm according to WHO methods . The sperm abnormality was evaluated according to the standard method of Narayana .Briefly, smears of the sperm suspension were made on clean glass slides and stained with periodic acid-Schiff's reaction haematoxylin. The stained smears were observed under a light microscopic with 40× magnification. The sperms were classified into normal and abnormal. The total sperm abnormality was expressed as percentage incidence. Other biochemical tests will be doing according the our research protocol and thesis for blood samples for measure LH, Testosterone, TAC, Glc and Cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* all patients suffering from oligospermia are included

Exclusion Criteria:

* any diseases

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Sperm count variation | First day of research, 2th time for sampling is 180 days after treatment
  Semen analysis according WHO methods

SECONDARY OUTCOMES:
Sperm motility | 1th time in first day of research, 2th time after 180 days of treatment
  Semen analysis
Sperm Viability | 1th time in first day of research, 2th time after 180 days of treatment
  Semen analysis

OTHER OUTCOMES:
Testosterone levels | 1th time in first day of research, 2th time after 180 days of treatment
  Testosterone analysis
Serum Total antioxidant levels | 1th time in first day of research, 2th time after 180 days of treatment
  Total antioxidant measurement in serum

CONTACTS AND LOCATIONS:
Overall Officials: Arash Khaki, PhD, Study Director — Women Reproductive Health Research Center,Tabriz University of medical Sciences
Locations (1):
- Womens Reproductive Health Research Center,Tabriz University Of Medical Sciences,Iran, Tabriz, Azarbyjan, Iran